CLINICAL TRIAL: NCT04189510
Title: Use of Closed Loop Insulin Delivery in the Immediate Postoperative Period Following Deceased Donor Kidney Transplant in Patients With Insulin Dependent Diabetes Mellitus
Brief Title: Use of Closed Loop Insulin Delivery for Glucose Control in Patients With Insulin Dependent Diabetes Mellitus After Kidney Transplantation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: ongoing concern of working with high-risk in-hospital transplant population during the various stages of the COVID-19 Pandemic.
Sponsor: University of Virginia (Other)
Collaborators: DexCom, Inc. (Industry); Tandem Diabetes Care, Inc. (Industry)
Responsible Party: Principal Investigator, Meaghan Stumpf, MD, Associate Professor, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 190055
Record Dates: First submitted 2019-11-22; First posted 2019-12-06 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Type 1 Diabetes; Insulin-requiring Type 2 Diabetes Mellitus; End Stage Renal Disease (ESRD)
Keywords: Type 1 Diabetes; Type 2 Diabetes; Artificial Pancreas (AP); Continuous Glucose Monitor (CGM); Kidney Transplant; Multiple Daily Injections (MDI)
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Kidney Failure, Chronic; Diabetes Mellitus, Type 2 | interventions — Pancreas, Artificial

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Artificial Pancreas (AP) Insulin Group (Experimental)
  Interventions: Device: Artificial Pancreas
- Multiple Daily Injections (MDI) Insulin Group (Active Comparator)
  Interventions: Other: Multiple Daily Injections

INTERVENTIONS:
Device: Artificial Pancreas — The Artificial Pancreas will delivery insulin in place of Multiple Daily Injections after a kidney transplant.
  Arms: Artificial Pancreas (AP) Insulin Group
Other: Multiple Daily Injections — Multiple Daily Injections as standard of care post kidney transplant.
  Arms: Multiple Daily Injections (MDI) Insulin Group

SUMMARY:
This study will be a prospective, single center, randomized controlled parallel group open-label trial. Participants with insulin requiring diabetes mellitus who have been offered an organ for living or deceased donor kidney transplantation will be recruited prior to transplantation surgery. Patients will be randomized in a 2:1 fashion to AP (6 patients) and conventional treatment groups (3 patients). At the end of the subject's post-operative in-patient stay, participants will have the option of wearing a blinded CGM at home for 4 weeks while treating themselves with multiple daily injections (MDI).

DETAILED DESCRIPTION:
The purpose of this study is to conduct a hypothesis-generating pilot study to assess the efficacy and safety of the closed loop control in kidney transplant recipients with history of insulin requiring diabetes mellitus in the early postoperative period.

This study will be a prospective, single center, randomized controlled parallel group open-label trial. Participants with insulin requiring diabetes mellitus who have been offered an organ for living or deceased donor kidney transplantation will be recruited prior to transplantation surgery. Patients will be randomized in a 2:1 fashion to AP (6 patients) and conventional treatment groups (3 patients). At the end of the subject's post-operative in-patient stay, participants will have the option of wearing a blinded CGM at home for 12 weeks while treating themselves with multiple daily injections (MDI).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18.0 years old at time of consent
2. History of insulin requiring diabetes mellitus, type 1 or type 2, who have end stage renal disease (ESRD)
3. Expected to undergo deceased or living donor kidney transplant surgery
4. History of insulin prescription (past or current use)
5. If female and sexually active, must agree to use a form of contraception to prevent pregnancy while a participant in the study. A negative serum or urine pregnancy test will be required for all females of childbearing potential. Participants who become pregnant will be discontinued from the study.
6. Willingness to switch to lispro (Humalog) or aspart (Novolog) if not using already, and to use no other insulin besides lispro (Humalog) or aspart (Novolog) during the study
7. Total daily insulin dose (TDD) at least 10 U/day
8. An understanding and willingness to follow the protocol and signed informed consent

Exclusion Criteria:

1. Pregnancy or intent to become pregnant during the trial
2. Currently breastfeeding or planning to breastfeed
3. A known medical condition that in the judgment of the investigator might interfere with the completion of the protocol.
4. Having a family member(s) employed by Tandem Diabetes Care, Inc. or having a direct supervisor at place of employment who is also directly involved in conducting the clinical trial (as a study investigator, coordinator, etc.); or having a first-degree relative who is directly involved in conducting the clinical trial.
5. Patients who have consented to participate in other interventional trials will be excluded or given the opportunity to exit from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety of Artificial Pancreas system | 5 Weeks
  Safety will be assessed by using a continuous glucose monitor, which measures interstitial glucose concentrations every 5 minutes for 24 hours a day. We will measure percentage of time in 24 hour period that the continuous glucose monitor (CGM) measures interstitial glucose values <70 mg/dL per day as a surrogate assessment of safety.
Efficacy of Artificial Pancreas system | 5 Weeks
  Efficacy will be assessed by using a continuous glucose monitor, which measures interstitial glucose concentrations every 5 minutes, 24 hours per day. We will measure percentage of time in 24 hour period that the continuous glucose monitor (CGM) measures interstitial glucose values between 70-180 mg/dL as a surrogate assessment of efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Meaghan Stumpf, MD, Principal Investigator — University of Virginia

IPD SHARING:
Plan to Share IPD: Undecided
Pending